CLINICAL TRIAL: NCT06426082
Title: Deciphering the Molecular and Secretory Functions of a Novel and Unique Brown Adipose Tissue Depot in Women
Brief Title: Deciphering a Novel and Unique Brown Adipose Tissue Depot in Women
Acronym: DEBATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Leiden University Medical Center (Other); ETH Zurich (Switzerland) (Other)
Responsible Party: Principal Investigator, Borja Martínez Tellez, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PID2022-141442OA-I00
Record Dates: First submitted 2023-10-11; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Cardiometabolic Diseases
Keywords: brown adipose tissue; cold exposure; hot exposure; dorsocervical fat; exercise
MeSH Terms: conditions — Motor Activity | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: This study will consist of a randomized controlled trial in which forty young, lean women will be assigned to a control group (n=10; receiving a thermoneutral exposure 2 hours/day at 32ºC; 5 days/week) or a cold exposure group (n=10; receiving 2 hours/day at 18ºC; 5 days/week) or aerobic exercise group (n=10; receiving 5 days/week at 65% heart rate reserve for 60 minutes each training session) or an ADBR2 agonist ingestion (n=10; salbutamol 12 mg/day. 7 days week).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Thermoneutral condition (Placebo Comparator): n=10; receiving a thermoneutral exposure 2 hours/day at 32ºC; 5 days/week; Total 4 weeks
  Interventions: Behavioral: Thermoneutral condition
- Cold condition (Experimental): n=10; receiving 2 hours/day at 18ºC; 5 days/week; Total 4 weeks
  Interventions: Behavioral: Cold condition
- Salbutamol (Experimental): n=10; salbutamol 12 mg/day. 7 days week. Total 4 weeks
  Interventions: Drug: Salbutamol
- Aerobic exercise (Experimental): n=10; receiving 5 days/week at 65% heart rate reserve for 60 minutes each training session. Total 4 weeks
  Interventions: Behavioral: Aerobic exercise condition

INTERVENTIONS:
Behavioral: Thermoneutral condition — Participants will be exposed 2 hours/day at 32ºC for 5 days/week
  Arms: Thermoneutral condition
Behavioral: Cold condition — Participants will be exposed 2 hours/day at 18ºC for 5 days/week
  Arms: Cold condition
Behavioral: Aerobic exercise condition — Participants will perform aerobic exercise training 5 days/week at 65% heart rate reserve for 60 minutes each training session
  Arms: Aerobic exercise
Drug: Salbutamol — Participants will take salbutamol 12 mg/day. 7 days week
  Arms: Salbutamol

SUMMARY:
Type of Study: Clinical Trial

Goal: The goal of this clinical trial is to investigate specific brown and beige fat cells in the dorsocervical area of young, lean adult women.

Participant Population/Health Conditions: The study will involve 40 young, lean adult women.

Main Questions: The main questions this study aims to answer are:

* Are there active brown or beige adipocytes in the subcutaneous fat of the dorsocervical area (i.e., iBAT)?
* What is the secretory function of these adipocytes?
* How do traditional interventions like cold exposure, as well as new approaches like Beta-2 agonist stimulation and exercise, affect the thermogenesis of these fat cells at the cellular and molecular levels?

Participants Will:

Be randomized into one of four groups: thermoneutral exposure, cold exposure, aerobic exercise, or Beta-2 agonist treatment.

Follow their assigned regimen for 4 weeks. Provide tissue samples from the dorsocervical area and abdomen before and after the 4-week intervention.

Undergo analysis of these samples using advanced techniques to understand the presence and activity of brown and beige fat cells.

Comparison Group: Researchers will compare the effects of different interventions (thermoneutral exposure, cold exposure, aerobic exercise, Beta-2 agonist treatment) on the presence and thermogenesis of brown and beige fat cells in the dorsocervical area.

DETAILED DESCRIPTION:
Cardiometabolic diseases affect almost 50% of the population in the Western World. While lifestyle plus pharmacological interventions may provide short-term benefits, more research is needed to understand the long-term effectiveness and underlying molecular mechanisms. Brown adipose tissue (BAT) is a thermogenic tissue that combusts large amounts of glucose and lipids to generate heat and secretes signalling molecules known as 'batokines' that can influence cardiometabolic health. Previous research has shown that BAT is active in adults, primarily in the supraclavicular region, as demonstrated by the uptake of 18F-Fluorodeoxyglucose. Recently, it has been demonstrated that a rare subpopulation of brown adipocytes increases their abundance at higher temperatures and can regulate the thermogenesis of neighbouring adipocytes. Thus, it is plausible that classical (e.g., cold exposure) and novel interventions (i.e., Beta-2 stimulation and exercise) that can activate BAT, would induce a remodelling in the brown/beige subpopulation adipocytes that govern whole tissue thermogenesis. These unstudied changes in human BAT physiology could potentially explain how BAT activation could enhance cardiometabolic health. However, despite over a decade of research, our understanding of the role of BAT in human physiology in humans is limited. This lack of knowledge may be mainly explained because i) obtaining biological samples of human BAT is very difficult and ii) the seasonal variation strongly influences the current gold standard (PET-CT scan). Given the pilot data found in this proposal, young, lean adult women may have a novel and undescribed thermogenic active BAT depot at the dorsocervical area (i.e., interscapular BAT=iBAT).

Based on that, the main hypothesis is that there are brown and/or beige adipocytes present within the subcutaneous adipose tissue of the dorsocervical area (i.e., iBAT) that have a unique composition of adipocyte subpopulations and specific secretory functions. Additionally, the specific subpopulations of brown and/or beige adipocytes related to thermogenesis in iBAT can be increased through exposure to cold temperatures, Beta-2 agonist stimulation, and exercise in young, lean women.

Thus, the main objective of this study is to investigate whether the subcutaneous fat in the dorsocervical area contains active brown and/or beige adipocytes (i.e., iBAT), understand its secretory function, and study the impact of traditional (e.g. cold exposure) and new interventions (e.g. Beta-2 agonist and exercise) on iBAT thermogenesis at the cellular and molecular levels.

Thus, the DEBATE project will carry out a randomized controlled trial where 40 young, lean adult women will be randomized into a thermoneutral exposure group (2 hours/day at 32ºC; 5 days/week) or a cold exposure group (2 hours/day at 18ºC; 5 days/week) or an aerobic exercise group (5 days/week at 65% heart rate reserve for 60 minutes) or a Beta-2 agonist group (salbutamol 12 mg/day. 7 days week). Before and after the 4-week intervention, iBAT tissue samples from the dorsocervical area and subcutaneous white adipose tissue (scWAT) from the abdomen will be collected. In these biological samples, the investigators will apply a set of cutting-edge omics (e.g., single nucleus RNA-seq) that will allow us to investigate whether iBAT is present and metabolically active in adults. The investigators will also conduct a set of in vitro experiments to discover the secretory function of this novel depot.

ELIGIBILITY:
Inclusion Criteria:

* 18-22 years of age women.
* BMI between ≥18 and <25 kg/m2
* Are willing to be randomized to either of these 4 groups.
* Must be sedentary (i.e., do not perform exercise or go to the gym).
* Participants should have regular menstrual cycles.
* Must be willing to adhere to all study procedures, including attendance at all study visits.
* Must be willing to have biological samples stored for future research.
* Must accept the use of the Period Calendar and Google Fit Apps on their mobile phones.

Exclusion Criteria:

* Diabetes mellitus (determined based on fasting glucose levels defined by ADA criteria).
* Any other active endocrine disease (thyroid disease, any signs of Cushing's syndrome, adrenal disease and lipid-associated disorders such as familial hypercholesterolemia).
* Any cardiac disease (i.e., ischemic cardiac disease, arrhythmias, severe heart failure).
* Use of medication known to influence glucose and/or lipid metabolism or brown fat activity (e.g., beta-blockers, antidepressants, corticosteroids).
* Use of medication shown to increase risk of hypokalemia after salbutamol administration (e.g., xanthine derivatives, steroids and diuretics).
* Clinically relevant abnormalities in clinical chemistry or electrocardiogram (ECG) at screening (to be judged by the study physician).
* A first-degree family member with sudden cardiac death.
* Any chronic renal or hepatic disease.
* Any other contra-indications for the use of salbutamol or propranolol.
* Abuse of alcohol or other substances.
* Smoking.
* Current participation in another research projects that may influence the current research project.
* Use of beta-adrenergic receptor agonists (e.g., asthma).
* Polycystic ovary syndrome.
* Diagnosed psychotic conditions.

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in UCP1 expression in the dorsocervical area | 2 years
  Investigators will quantify the level UCP1 expression by qPCR in white adipose tissue biopsies obtained before and after the intervention

SECONDARY OUTCOMES:
Body composition (BIA, Tanita) | 2 years
  Change in fat percentage (% of fat)
Cardiorespiratory fitness test (indirect calorimetry and monarch bike) | 2 years
  Change in VO2max (ml/kg/min)
LDL quantification in blood | 2 years
  Change in LDL-C (mg/dL)
HDL quantification in blood | 2 years
  Change in HDL-C (mg/dL)
Glucose quantification in blood | 2 years
  Change in Glucose (mg/dL)
Insulin quantification in blood | 2 years
  Change in Insulin (µIU/mL)
Triglycerides quantification in blood | 2 years
  Change in Triglycerides (mg/dL)
C-reactive protein quantification in blood | 2 years
  Change in CRP (mg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 5 years after publishing the data
Access Criteria: Everybody
URL: https://www.sportresearchgroup.es/

REFERENCES:
- [Background] Martinez-Tellez B, Sanchez-Delgado G, Alcantara JMA, Acosta FM, Amaro-Gahete FJ, Osuna-Prieto FJ, Perez-Bey A, Jimenez-Pavon D, Llamas-Elvira JM, Gil A, Aguilera CM, Rensen PCN, Ruiz JR. Evidence of high 18 F-fluorodeoxyglucose uptake in the subcutaneous adipose tissue of the dorsocervical area in young adults. Exp Physiol. 2019 Feb;104(2):168-173. doi: 10.1113/EP087428. Epub 2018 Dec 18. PMID 30468689